CLINICAL TRIAL: NCT04990245
Title: APOLLO Study: pAtient rePorted Outcomes Linked With histoLogy in Patients With uLcerative cOlitis
Brief Title: pAtient rePorted Outcomes Linked With histoLogy in Patients With uLcerative cOlitis
Acronym: APOLLO
Status: Completed | Type: Observational
Sponsor: Imelda GI Clinical Research Center (Other)
Responsible Party: Sponsor
Other Study IDs: 200735
Record Dates: First submitted 2021-07-29; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; patient reported outcomes; histological scoring; disability; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — intestinale biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ulcerative colitis: patients with ulcerative colitis and planned endoscopy as part of routine care
  Interventions: Diagnostic Test: endoscopic biopsies

INTERVENTIONS:
Diagnostic Test: endoscopic biopsies — patients with planned endoscopy for ulcerative colitis have endosocpic data recorded aswell as biopsy sampling and blood tests

SUMMARY:
Background and rationale:

In ulcerative colitis, treating beyond endoscopic healing has shown a reduction of relapse and hospitalization, pushing for histological remission in daily clinical practice.1 However, very little is known on how histological remission is associated with patient reported outcomes (PROMs).2,3 In recent years, several questionnaires have been developed to assess what really matters to patients: symptoms and the burden UC exerts on them.4 As PROMs are getting more and more attention during drug development programs and drug approval by international organizations, including FDA and EMA, the link between objective outcome measures (endoscopic, histological, biochemical) and PROMs should therefore be better characterized.

Objectives and design:

To investigate prospectively the association of patient reported outcomes (PROMs) and biochemical, endoscopic and histological outcome measures in patients with ulcerative colitis.

DETAILED DESCRIPTION:
After informed consent, patients will undergo endoscopic assessment evaluating endoscopic disease activity using established scoring systems

* Mayo endoscopic sub-score5
* Ulcerative Colitis Endoscopic Index of Severity [UCEIS]6 All endoscopic assessments will be recorded, allowing blinded scoring by independent endoscopists afterwards. Study protocol APOLLO - 2 During endoscopy, colonic biopsies will be taken according to standard of care from the most inflamed area of the colon and normal area if applicable, 0-60cm from the anal verge. All biopsies will be scored histologically using the Nancy Index.7 During the same study visit, clinical symptoms (Simple clinical colitis activity index [SCCAI]) and patient reported outcomes (PROMs) will be evaluated digitally using validated scoring systems8
* IBD disk
* PRO-2
* Visual Analogue Scale
* IBD control in case of non-remission Finally, patients will be biochemically (C-reactive protein, hemoglobin, albumin) evaluated, including measurement of drug level (infliximab, adalimumab, vedolizumab) in case of ongoing exposure to biological agents. All evaluations are part of standard-of-care. Definitions
* Endoscopic remission: Mayo endoscopic sub-score 0 AND UCEIS 0
* Endoscopic response according to

  * Mayo score: decrease in Mayo endoscopic sub-score ≥ 1
  * UCEIS: decrease in UCEIS ≥ 2
* Endoscopic improvement: Mayo endoscopic sub-score 1
* Histological remission: Nancy histological index 0
* Absence of active/acute histological inflammation: Nancy histological index 0-1
* Histological response: Nancy histological index > 1
* PRO2 remission: stool frequency ≤ 1 (absolute stool frequency ≤ 3 OR 1-2 stools more than usual) AND rectal bleeding score of 0 (average of 3 days prior to endoscopy)
* IBD disk remission per item:

  * Abdominal pain
  * Regulating defecation
  * Interpersonal interactions
  * Education and work
  * Sleep
  * Energy
  * Emotions
  * Body Image
  * Sexual function
  * Joint pain

ELIGIBILITY:
INCLUSION CRITERIA:

All patients with ulcerative colitis (≥ 16 years) undergoing planned endoscopic assessment as part of standard of care between 01.07.2020 and 30.06.2021. Evidence of a personally signed and dated informed consent document (ICF) indicating that the subject has been informed of all aspects of the study.

EXCLUSION CRITERIA:

Subjects with a diagnosis of indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, microscopic colitis or Crohn's disease.

Subjects with clinical findings suggestive of CD (e.g. fistulae, granulomas on biopsy) are also excluded. Similar data collection within 8 weeks prior to endoscopic assessment

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with ulcerative colitis and planned endoscopy as part of routine care
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
correlation between histological disease activity and disability | 1 day
  histological activity is based on the Nancy score, disability is based on the IBD disk

SECONDARY OUTCOMES:
correlation between histological disease activity and patient reported outcomes | 1 day
  histological activity is based on the Nancy score, PRO is based on the SCCAI
correlation between histological disease activity and patient reported outcomes | 1 day
  histological activity is based on the Nancy score, PRO is based on the VAS
correlation between histological disease activity and patient reported outcomes | 1 day
  histological activity is based on the Nancy score, PRO is based on the PRO-2
correlation between histological disease activity and endoscopic disease activity | 1 day
  histological activity is based on the Nancy score, endoscopic disease activityis based on the Mayo endoscopic subscore
correlation between histological disease activity and endoscopic disease activity | 1 day
  histological activity is based on the Nancy score, endoscopic disease activity is based on the UCEIS
correlation between histological disease activity and biomarkers | 1 day
  histological activity is based on the Nancy score, biomarkers (CRP, hemoglobine, albumin)

OTHER OUTCOMES:
correlation between histological disease activity and patient reported outcomes | 1 day
  histological activity is based on the Nancy score, disability is based on the IBD control in case of non remission

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bossuyt, MD, Principal Investigator — Imelda general hospital
Locations (1):
- Imelda GI clinical research center, Bonheiden, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
up on request

REFERENCES:
- [Background] Danese S, Roda G, Peyrin-Biroulet L. Evolving therapeutic goals in ulcerative colitis: towards disease clearance. Nat Rev Gastroenterol Hepatol. 2020 Jan;17(1):1-2. doi: 10.1038/s41575-019-0211-1. No abstract available. PMID 31520081
- [Background] Colombel JF, Keir ME, Scherl A, Zhao R, de Hertogh G, Faubion WA, Lu TT. Discrepancies between patient-reported outcomes, and endoscopic and histological appearance in UC. Gut. 2017 Dec;66(12):2063-2068. doi: 10.1136/gutjnl-2016-312307. Epub 2016 Sep 2. PMID 27590995
- [Background] Dragasevic S, Sokic-Milutinovic A, Stojkovic Lalosevic M, Milovanovic T, Djuranovic S, Jovanovic I, Rajic S, Stojkovic M, Milicic B, Kmezic S, Oluic B, Aleksic M, Pavlovic Markovic A, Popovic D. Correlation of Patient-Reported Outcome (PRO-2) with Endoscopic and Histological Features in Ulcerative Colitis and Crohn's Disease Patients. Gastroenterol Res Pract. 2020 Apr 2;2020:2065383. doi: 10.1155/2020/2065383. eCollection 2020. PMID 32328091
- [Background] de Jong MJ, Huibregtse R, Masclee AAM, Jonkers DMAE, Pierik MJ. Patient-Reported Outcome Measures for Use in Clinical Trials and Clinical Practice in Inflammatory Bowel Diseases: A Systematic Review. Clin Gastroenterol Hepatol. 2018 May;16(5):648-663.e3. doi: 10.1016/j.cgh.2017.10.019. Epub 2017 Oct 23. PMID 29074448
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Travis SP, Schnell D, Krzeski P, Abreu MT, Altman DG, Colombel JF, Feagan BG, Hanauer SB, Lichtenstein GR, Marteau PR, Reinisch W, Sands BE, Yacyshyn BR, Schnell P, Bernhardt CA, Mary JY, Sandborn WJ. Reliability and initial validation of the ulcerative colitis endoscopic index of severity. Gastroenterology. 2013 Nov;145(5):987-95. doi: 10.1053/j.gastro.2013.07.024. Epub 2013 Jul 25. PMID 23891974
- [Background] Marchal-Bressenot A, Salleron J, Boulagnon-Rombi C, Bastien C, Cahn V, Cadiot G, Diebold MD, Danese S, Reinisch W, Schreiber S, Travis S, Peyrin-Biroulet L. Development and validation of the Nancy histological index for UC. Gut. 2017 Jan;66(1):43-49. doi: 10.1136/gutjnl-2015-310187. Epub 2015 Oct 13. PMID 26464414
- [Background] Bossuyt P, Hoefkens E, Pouillon L. Prime Time Was Yesterday for Patient-reported Outcomes in Daily Care of Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2018 Nov;16(11):1839. doi: 10.1016/j.cgh.2018.05.029. No abstract available. PMID 30343866